CLINICAL TRIAL: NCT01087723
Title: Multi-centre, Multi-national, Prospective, Randomised, Open-label, Comparison of Bivalirudin to Other Guideline Based Current Therapies (Excluding Bivalirudin)
Brief Title: European Ambulance Acute Coronary Syndrome (ACS) Angiography Trial
Acronym: EUROMAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-08-03
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome
Keywords: EUROMAX; STEMI; STE-ACS; UFH; bivalirudin; PCI; ambulance study; STE-MI participants
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction | interventions — bivalirudin; Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalirudin (Experimental): Given immediately upon enrollment as an intravenous (IV) bolus of 0.75 mg/kilogram (mg/kg), followed immediately by an infusion of 1.75 mg/kg/hour (mg/kg/h). This infusion was to be run continuously until completion of PCI, at which time the infusion was reduced to 0.25 mg/kg/h for at least 4 hours. An optional PCI-dose infusion of 1.75 mg/kg/h was also permitted for up to 4 hours at the discretion of the operator.
  Interventions: Drug: Bivalirudin
- Standard of Care: Heparins with Optional GPI (Active Comparator): Standard-of-care anti-thrombotic therapy as outlined in the European Society of Cardiology Dosing Guidelines for Management of STE-ACS, not including bivalirudin: UFH (100 international units/kg [IU/kg] without GPI and 60 IU/kg with GPI). Any of the following approved GPIs were used either as a routine strategy or as a bail out: eptifibatide (two 180-micrograms/kilogram [μg/kg] IV boluses with a 10-minute [min] interval followed by an infusion of 2.0 μg/kg/min for 72-96 hours); tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18-24 hours); or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours [maximum dose of 10 μg/min]).
  For this study, the control consisted of treatment with UFH or low molecular weight heparin (LMWH) with or without GPI and is referred to as "heparins with optional GPI."
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin
  Other Names: Angiox; Angiomax
  Arms: Bivalirudin
Drug: Heparin
  Other Names: UFH; LMWH
  Arms: Standard of Care: Heparins with Optional GPI

SUMMARY:
To show that the early administration of bivalirudin improves 30 day outcomes when compared to the current standard of care in participants with ST segment elevation acute coronary syndrome (STE-ACS), intended for a primary percutaneous coronary intervention (PCI) management strategy, presenting either via ambulance or to centers where PCI is not performed.

DETAILED DESCRIPTION:
The purpose of the trial is to show that the early administration of bivalirudin improves 30-day outcomes when compared to the current standard of care in participants with STE-ACS, with an onset of symptoms of >20 minutes and <12 hours, intended for a primary PCI management strategy, presenting either via ambulance or to centers where PCI is not performed.

All participants are to receive treatment with aspirin (150-325 milligrams [mg] administered orally or 250-500 mg intravenously [IV]), followed by 75-100 milligrams/day (mg/day) for at least 1 year and a loading dose of an approved P2Y12 receptor blocker, such as clopidogrel, prasugrel, or ticagrelor, that was to be continued as per European Society of Cardiology guidelines (preferably for 1 year) in all participants.

The primary objectives of the trial are to show that, when compared with standard anti-thrombotic therapies other than bivalirudin (which includes treatment with unfractionated heparin [UFH] and optional glycoprotein IIb/IIIa inhibitor [GPI]) that at 30 days:

• Bivalirudin is superior to control at reducing a composite of death and non-coronary artery bypass graft (CABG)-related protocol major bleeding.

ELIGIBILITY:
Inclusion Criteria:

The decision to randomize participants was made by a qualified physician or paramedic who was present at the time.

Participants were included in the study if they presented either via ambulance or to a center where PCI was not performed and met all of the following criteria:

1. Provided written informed consent before initiation of any study related procedures. Participants randomized in the ambulance may initially have signed an abridged version.
2. Aged ≥18 years at the time of randomization.
3. Had a presumed diagnosis of STE-ACS with onset of symptoms of >20 minutes and <12 hours with one or more of the following:

   * ST segment elevation of ≥1 millimeters (mm) in ≥2 contiguous leads
   * Presumably new left bundle branch block
   * An infero-lateral myocardial infarction with ST segment depression of ≥1 mm in ≥2 of leads V1-3 with a positive terminal T wave
4. All participants would proceed with emergent angiography and primary PCI if indicated <2 hours after first medical contact

Exclusion Criteria:

Participants were excluded from the study if any of the following exclusion criteria applied prior to randomization:

1. Any bleeding diathesis or severe hematological disease or history of intra-cerebral mass, aneurysm, arterio-venous malformation, hemorrhagic stroke, intra-cranial hemorrhage, or gastrointestinal or genitourinary bleeding within the last 2 weeks.
2. Participants who had undergone recent surgery (including biopsy) within the last 2 weeks.
3. Participants who were on warfarin (not applicable if International Normalized Ratio known to be <1.5).
4. Participants who had received UFH, LMWH, or bivalirudin immediately before randomization.
5. Thrombolytic therapy within the last 48 hours.
6. Absolute contra-indications or allergy that could not be pre-medicated to iodinated contrast or to any of the study medications including aspirin or clopidogrel.
7. Contraindications to angiography, including but not limited to severe peripheral vascular disease.
8. If it was known, pregnant or nursing mothers. Women of child-bearing age were asked if they were pregnant or thought that they may be pregnant.
9. If it is known, a creatinine clearance <30 milliliter/minute or dialysis dependent.
10. Previous enrolment in this study.
11. Treatment with other investigational drugs or devices within the 30 days preceding randomization or planned use of other investigational drugs or devices in this trial.
12. Participants may not have been enrolled if the duration of randomized investigational medicinal product anti-thrombin infusion was likely to be <30 minutes from the time of onset to the commencement of angiography.
13. Participants may not have been enrolled within a primary PCI-capable hospital (unless at the time of randomization, the catheter laboratory was not available, and the participant required transfer to another primary PCI capable hospital).
14. Estimated body weight of >120 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2198 (Actual)
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Steg, Prof, Study Chair — Executive Committee; Christian Hamm, BSc, MD, PhD, Study Chair — International Steering Committee
Locations (145):
- Austria (4):
  - Hanusch Krankenhaus, Vienna
  - Magistratsabeilung 70, Wiener, Vienna
  - Universitats-Klinik Fur, Vienna
  - Wilhelminenspital MA 6 - BA 19, Vienna
- Zdravotnicka Zachranna Sluzba, České Budějovice, Czechia
- Denmark (7):
  - Aarhus Universitetshospital, Aarhus
  - Akutlaegebil Kobenhavn, Hc Andersens Boulevard 23, Copenhagen
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Hellerup
  - Akutlaegebil Nordsjaelland, Hillerød
  - Laegeambulancen Odense, Odense
  - Odense Universitets Hospital, Odense
- France (44):
  - Hopital Europeen Paris La Roseraie, Aubervilliers
  - Hospital Avicenne, Pharmacie -Gestion Des Essais Cliniques, Bobigny
  - Chu De Bordeaux - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Bourg En Bresse, Bourg-en-Bresse
  - Clinique Convert, Bourg-en-Bresse
  - Ch Jacques Coeur, Bourges
  - Centre Hospitalier Universitaire De Caen, Caen
  - Hopital Prive Saint Martin, Caen
  - Service De Cardiologie, Cedex
  - Ch Chateauroux, Châteauroux
  - Chu Clermont-Ferrand, Hopital, Clermont-Ferrand
  - Samu-Smur Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Ch Sud Francilien - Site Corbeil, Corbeil Essonne
  - Ch Sud Francilien - Site Corbeil, Pharmacie, Corbeil-Essonnes
  - Capio - Clinique Des Cedres, Cornebarrieu
  - Hospital Henri Mondor, Pharmacie, Créteil
  - Samu 92 Hauts De Seine, Garches
  - Clinique Les Eaux Claires Ghm, Grenoble
  - Chu A Michallon Grenoble, La Tronche
  - Samu Chu A Michallon Grenoble, La Tronche
  - Hopital Andre Mignot - Centre Hospitalier De Versailles, Le Chesnay
  - Chr Lille, Lille
  - Samu 59/Samu Du Nord, Lille
  - Centre Hospitalier De Longjumeau, Longjumeau
  - Centre Hospitalier St Joseph St Luc, Lyon
  - Institut Hospitalier Jacques Cartier, Massy
  - Centre Hospitalier De Montelimar, Montélimar
  - Chi Le Raincy - Montfermeil Site De Montfermeil, Montfermeil
  - Clinique Ambroise Pare, Neuilly
  - Centre Hospitalier, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Ch De Pau Hopital Francois Mitterand, Pau
  - Samu Ch De Pau, Pau
  - Cardiologic Hospital - Coronary Care Unit, University of Bordeaux, Pessac
  - Clinique Belledonne, Saint-Martin-d'Hères
  - Pole Smur, Samu 77 - Medecine, Seine Et Marne
  - Chu De Toulouse - Hopital Paule De Viguier, Toulouse
  - Chu Toulouse - Hopital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Polyclinique Du Parc, Toulouse
  - Centre Hospitalier De Valence, Valence
  - Centre Hospitalier De Vienne Centre Hospitalier Lucien Hussel, Vienne
- Germany (16):
  - Kerckhoff Heart Center, Bad Nauheim
  - Rettungsdienst Wetteraukreis, Bad Nauheim
  - Charite Universitatsmedizin Berlin Campus Virchow-Klinikum, Berlin
  - Lutzowstrabe, Berlin
  - Sana Klinikum Lichtenberg Oskar Ziethen Krankenhaus, Fanningerstrasse 32, Berlin
  - Universitatsklinikum Benjamin Franklin, Hindenburgdamm 30, Berlin
  - Klinikum Links Der Weser, Bremen
  - Evangelisches Bethesda Johanniter, Duisburg
  - Feuerwehr Duisburg, Duisburg
  - Herzzentrum Duisburg, Klinik Fur Kardiologie And Angiologie, Duisburg
  - Klinikum Duisburg Ggmbh, Duisburg
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt
  - Medizinische Hochschule Hannover, Carl Neuberg Str. 1, Hanover
  - Klinikum Ludwigshafen, Ludwigshafen
  - Stadtisches Klinikum Luneburg, Bogelstr. 1, Lüneburg
  - Helios Klinik Der Universitat Witten Herdecke, Wuppertal
- Italy (10):
  - Ospedale Maggiore, Bologna
  - Ospedle Di Bentivoglio, Bologna
  - Policlinico S.Orsola Malpighi, Bologna
  - Ospedale Di Assisi, Perugia
  - Ospedale Di Castiglione Del Lago, Perugia
  - Ospedale Di Todi, Perugia
  - Ospedale S.Maria Misericordia, Perugia
  - Asur Marche- Zona 1 Pesaro, Pesaro
  - Azienda Ospedaliera San Salvatore, Pesaro
  - Emergency Rescue & Mobile Als Unit, Lanciarini Pub, Pesaro
- Netherlands (17):
  - Betreft Research Regional, Amersfoort
  - Meander Medisch Centrum, Amersfoort
  - Rav Noord En Oost Gelderland, Amersfoort
  - Pharmacy Department, Nieuwegein
  - Regional Ambulance Service Gelderland Midden, Nieuwegein
  - St Antonius Ziekenhuis, Nieuwegein
  - Service Gelderland-Zuid Klinisch Geneesmiddelonderzoek Klinsche Farmacie Afd Klinsche Farmacie, Nijmegan
  - Cwz Klinisch Geneesmiddelonderzoek Klinische, Nijmegen
  - Kgo Team Regional Ambulance, Nijmegen
  - Regional Ambulance Service Gelderland Zuid, Nijmegen
  - Regional Ambulance Service Gelderland-Zuid Distributiecentrum, Nijmegen
  - Regional Ambulance Service, Nijmegen
  - Umc St.Radboud Nijmegen, Nijmegen
  - Department Of Cardiology, Utrecht
  - Umc Utrecht, Utrecht
  - Isala Klinieken, Zwolle
  - Tav Trial Team, Isala Klinieken Ioc Weezenlanden Afd, Zwolle
- Poland (32):
  - Poradnia Kardiologiczna, Będzin
  - Malopolskie Centrum Sercowo, Chrzanów
  - Szpital Powiatowy W Chrzanowie, Chrzanów
  - Oddzial Polskiej-Amerikanskiej Kliniki Serca, Dąbrowa Górnicza
  - Szpital Powiatowy W Debicy, Dębica
  - Specialist Hospital Gorlice, Gorlice
  - Szpital Powiatowy Im. Jana Pawla Ii W Kolbuszowej, Kolbuszowa
  - Jagiellonian University Medical College,, Krakow
  - Krakowskie Centrum, Krakow
  - Oddzial Kardiologii, Krakow
  - Samodzielny Publiczny Zaklad Opieki, Krakow
  - Szpital Specjalistyczny Im Szpitalny Oddzial Ratunkowy, Krakow
  - Spzoz Szpital Im. J.Dietla W Krynicy Zdroj, Krynica-Zdrój
  - Szpital Powiatowy W Limanowej, Limanowa
  - Szpital Bieganskiego, Lodz
  - Medical University Of Lublin, Lublin
  - Polsko-Amerykanskie Kliniki Serca, Szpital Powiatowy, Mielec
  - Samodzielny Pobliszny Zaklad W Mielcu, Mielec
  - Myslowickie Centrum Zdrowia, Mysłowice
  - Samodzielna Publiczna Stacja Pogotowia Ratunkowego, Samodzielna Publiczna Stacja Pogotowia Ratunkowego W Niepolomicach, Niepołomice
  - Intercard Nowy Sacz, Nowy Sącz
  - Nzoz Nowy Szpital W Olkuszu, Olkusz
  - Szpital Powiatowy, Opatów
  - Carint, Ostrowiec Świętokrzyski
  - Spzoz Parczew, Parczew
  - Samodzielny Szpital Wojewodski, Piotrkow Trybunalski
  - Spzoz W Radzyniu Podlaskim, Radzyń Podlaski
  - Szpital Powiatowy W Sedziszowie Malopolskim, Sędziszów Małopolski
  - Oddzial Chorob Wewnetrznych, Staszów
  - Oddzial Kardiologii Al.Lotnikow Polskich 18, Świdnik
  - Szpital Zakonu Bonifratrow Sw., Todz
  - Spzoz Lask, Łask
- Slovenia (14):
  - Zdravstveni Dom Celje, Celje
  - Splosna Bolnisnica Izola, Polje 40, Izola
  - Oe Zdravstveni Dom Jesenice, Jesenice
  - Splosna Bolnisnica Jesenic, Jesenice
  - Zdravstveni Dom Lenart, Maistrova 22, Lenart v Slov. Goricah
  - Univerzitetni Klinicni Center Ljubljana, Ljubljana
  - Zdravstveni Dom Ljubljana, Ljubljana
  - Univerzitetni Klinicni Center Maribor, Maribor
  - Zdravstveni Dom Dr. Adolfa Drolca Maribor, Maribor
  - Splosna Bolnisnica Novo Mesto/ Community Hospital Novo Mesto, Smihelska Cesta 1, Novo Mesto
  - Zdravstveni Dom Ormoz, Ormož
  - Splosna Bolnisnica Ptuj, Interni Odelek, Potrceva Cesta 23, Ptuj
  - Zdravstveni Dom Slovenska Bistrica, Slovenska Bistrica
  - Zdravstveni Dom Slovenske Konjice, Slovenske Konjice

REFERENCES:
- [Derived] Huber K, Ducrocq G, Hamm CW, van 't Hof A, Lapostolle F, Coste P, Gordini G, Steinmetz J, Verheugt FWA, Adgey J, Nibbe L, Kanic V, Clemmensen P, Zeymer U, Bernstein D, Prats J, Deliargyris EN, Gabriel Steg P. Early clinical outcomes as a function of use of newer oral P2Y12 inhibitors versus clopidogrel in the EUROMAX trial. Open Heart. 2017 Nov 28;4(2):e000677. doi: 10.1136/openhrt-2017-000677. eCollection 2017. PMID 29225903
- [Derived] Fabris E, Kilic S, Van't Hof AWJ, Ten Berg J, Ayesta A, Zeymer U, Hamon M, Soulat L, Bernstein D, Anthopoulos P, Deliargyris EN, Steg PG. One-Year Mortality for Bivalirudin vs Heparins Plus Optional Glycoprotein IIb/IIIa Inhibitor Treatment Started in the Ambulance for ST-Segment Elevation Myocardial Infarction: A Secondary Analysis of the EUROMAX Randomized Clinical Trial. JAMA Cardiol. 2017 Jul 1;2(7):791-796. doi: 10.1001/jamacardio.2016.5975. PMID 28273285
- [Derived] Ducrocq G, Steg PG, Van't Hof A, Zeymer U, Mehran R, Hamm CW, Bernstein D, Prats J, Deliargyris EN, Stone GW. Utility of post-procedural anticoagulation after primary PCI for STEMI: insights from a pooled analysis of the HORIZONS-AMI and EUROMAX trials. Eur Heart J Acute Cardiovasc Care. 2017 Oct;6(7):659-665. doi: 10.1177/2048872616650869. Epub 2016 Jun 10. PMID 27287251
- [Derived] Dangas GD, Schoos MM, Steg PG, Mehran R, Clemmensen P, van 't Hof A, Prats J, Bernstein D, Deliargyris EN, Stone GW. Early Stent Thrombosis and Mortality After Primary Percutaneous Coronary Intervention in ST-Segment-Elevation Myocardial Infarction: A Patient-Level Analysis of 2 Randomized Trials. Circ Cardiovasc Interv. 2016 May;9(5):e003272. doi: 10.1161/CIRCINTERVENTIONS.115.003272. PMID 27165710
- [Derived] Kilic S, Van't Hof AW, Ten Berg J, Lopez AA, Zeymer U, Hamon M, Soulat L, Bernstein D, Deliargyris EN, Steg PG. Frequency and prognostic significance of access site and non-access site bleeding and impact of choice of antithrombin therapy in patients undergoing primary percutaneous coronary intervention. The EUROMAX trial. Int J Cardiol. 2016 May 15;211:119-23. doi: 10.1016/j.ijcard.2016.02.131. Epub 2016 Mar 3. PMID 26995053
- [Derived] Hamon M, Coste P, Van't Hof A, Ten Berg J, Clemmensen P, Tabone X, Benamer H, Kristensen SD, Cavallini C, Marzocchi A, Hamm C, Kanic V, Bernstein D, Anthopoulos P, Deliargyris EN, Steg PG. Impact of arterial access site on outcomes after primary percutaneous coronary intervention: prespecified subgroup analysis from the EUROMAX trial. Circ Cardiovasc Interv. 2015 Jun;8(6):e002049. doi: 10.1161/CIRCINTERVENTIONS.114.002049. PMID 26056249
- [Derived] Stone GW, Mehran R, Goldstein P, Witzenbichler B, Van't Hof A, Guagliumi G, Hamm CW, Genereux P, Clemmensen P, Pocock SJ, Gersh BJ, Bernstein D, Deliargyris EN, Steg PG. Bivalirudin versus heparin with or without glycoprotein IIb/IIIa inhibitors in patients with STEMI undergoing primary percutaneous coronary intervention: pooled patient-level analysis from the HORIZONS-AMI and EUROMAX trials. J Am Coll Cardiol. 2015 Jan 6;65(1):27-38. doi: 10.1016/j.jacc.2014.10.029. PMID 25572507
- [Derived] Steg PG, van 't Hof A, Clemmensen P, Lapostolle F, Dudek D, Hamon M, Cavallini C, Gordini G, Huber K, Coste P, Thicoipe M, Nibbe L, Steinmetz J, Ten Berg J, Eggink GJ, Zeymer U, Campo dell' Orto M, Kanic V, Deliargyris EN, Day J, Schuette D, Hamm CW, Goldstein P. Design and methods of European Ambulance Acute Coronary Syndrome Angiography Trial (EUROMAX): an international randomized open-label ambulance trial of bivalirudin versus standard-of-care anticoagulation in patients with acute ST-segment-elevation myocardial infarction transferred for primary percutaneous coronary intervention. Am Heart J. 2013 Dec;166(6):960-967.e6. doi: 10.1016/j.ahj.2013.08.025. Epub 2013 Nov 7. PMID 24268209
- [Derived] Steg PG, van 't Hof A, Hamm CW, Clemmensen P, Lapostolle F, Coste P, Ten Berg J, Van Grunsven P, Eggink GJ, Nibbe L, Zeymer U, Campo dell' Orto M, Nef H, Steinmetz J, Soulat L, Huber K, Deliargyris EN, Bernstein D, Schuette D, Prats J, Clayton T, Pocock S, Hamon M, Goldstein P; EUROMAX Investigators. Bivalirudin started during emergency transport for primary PCI. N Engl J Med. 2013 Dec 5;369(23):2207-17. doi: 10.1056/NEJMoa1311096. Epub 2013 Oct 30. PMID 24171490

RESULTS

PARTICIPANT FLOW:
Groups:
- Bivalirudin: Given immediately upon enrolment as an intravenous (IV) bolus of 0.75 milligrams/kilogram (mg/kg), followed immediately by an infusion of 1.75 mg/kg/hour (mg/kg/h). This infusion was to be run continuously until completion of percutaneous coronary intervention (PCI), at which time the infusion was reduced to 0.25 mg/kg/h for at least 4 hours. An optional PCI-dose infusion of 1.75 mg/kg/h was also permitted for up to 4 hours at the discretion of the operator.
- Standard of Care: Heparins With Optional GPI: Standard-of-care anti-thrombotic therapy as outlined in the European Society of Cardiology Dosing Guidelines for Management of ST segment elevation acute coronary syndrome (STE-ACS ), not including bivalirudin: unfractionated heparin (UFH) (100 international units/kg [IU/kg] without glycoprotein IIb/IIIa inhibitor [GPI] and 60 IU/kg with GPI). Any of the following approved GPIs were used either as a routine strategy or as a bail out: eptifibatide (two 180-micrograms/kilogram [μg/kg] IV boluses with a 10-minute [min] interval followed by an infusion of 2.0 μg/kg/min for 72-96 hours); tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18-24 hours); or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours [maximum dose of 10 μg/min]).
  For this study, the control consisted of treatment with UFH or low molecular weight heparin (LMWH) with or without GPI and is referred to as "heparins with optional GPI."
Period: Overall Study
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Started | 1089 (Randomized participants who signed an informed consent form (ICF); Intent-to-treat (ITT) population) | 1109 (Randomized participants who signed an informed consent form (ICF); Intent-to-treat (ITT) population)
Received at Least 1 Dose of Study Drug | 1099 (Participants who were randomized with signed ICF by treatment actually received; Safety population) | 1094 (Participants who were randomized with signed ICF by treatment actually received; Safety population)
Completed | 1075 (Completed 1-year follow-up in the study) | 1089 (Completed 1-year follow-up in the study)
Not Completed | 14 | 20
Not completed — 1 Year Visit Too Early (<335 days) | 0 | 1
Not completed — Withdrawal by Subject | 10 | 13
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Reason Not Specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and signed an ICF; ITT population
Groups:
- Bivalirudin: Given immediately upon enrollment as an IV bolus of 0.75 mg/kg, followed immediately by an infusion of 1.75 mg/kg/h. This infusion was to be run continuously until completion of PCI, at which time the infusion was reduced to 0.25 mg/kg/h for at least 4 hours. An optional PCI-dose infusion of 1.75 mg/kg/h was also permitted for up to 4 hours at the discretion of the operator.
- Standard of Care: Heparins With Optional GPI: Standard-of-care anti-thrombotic therapy as outlined in the European Society of Cardiology Dosing Guidelines for Management of STE-ACS, not including bivalirudin: UFH (100 international IU/kg without GPI and 60 IU/kg with GPI). Any of the following approved GPIs were used either as a routine strategy or as a bail out: eptifibatide (two 180-μg/kg IV boluses with a 10-min interval followed by an infusion of 2.0 μg/kg/min for 72-96 hours); tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18-24 hours); or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours [maximum dose of 10 μg/min]).
  For this study, the control consisted of treatment with UFH or LMWH with or without GPI and is referred to as "heparins with optional GPI."
- Total: Total of all reporting groups
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI | Total
Number analyzed (Participants) | 1089 | 1109 | 2198
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (12.8) | 62.0 (13.1) | 61.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 248 | 523
  Male | 814 | 861 | 1675
Region of Enrollment [Number; unit: participants]
  Austria | 4 | 5 | 9
  Czech Republic | 0 | 1 | 1
  Netherlands | 377 | 391 | 768
  Denmark | 78 | 72 | 150
  Poland | 55 | 56 | 111
  Italy | 31 | 41 | 72
  France | 398 | 397 | 795
  Germany | 139 | 140 | 279
  Slovenia | 7 | 6 | 13
Medical history: Participant Has Diabetes [Number; unit: participants] | 127 | 169 | 296
Medical history: Participant Is a Current smoker (within past 30 days) [Number; unit: participants] | 453 | 472 | 925
Medical history: Participant Has Hypertension [Number; unit: participants] | 459 | 504 | 963
Medical history: Participant Has Hyperlipidemia [Number; unit: participants] — Participant has known hyperlipidemia or is on lipid-lowering drugs
  participants | 398 | 417 | 815
Medical history: Participant Has Had Previous myocardial infarction (MI) [Number; unit: participants] | 380 | 113 | 493

OUTCOME MEASURES:

1. Primary Outcome: The Composite Incidence of Death and Non-coronary Artery Bypass Graft (CABG) Major Bleeding
Description: A participant was defined to have had a composite event if the participant experienced at least 1 of the 2 components (death or non-CABG major bleeding) of the composite. Incidence=the number of participants to experience the event/total number of at risk participants x 100. Death was defined as death from any cause at any time. Non-CABG major bleeding was defined as any 1 of the following: intra-cranial, retroperitoneal, intraocular, access site hemorrhage requiring radiological or surgical intervention, reduction in hemoglobin (Hb) concentration of >4 grams/deciliter (g/dL) without an overt source of bleeding, reduction in hemoglobin concentration of >3 g/dL with an overt source of bleeding; re-intervention for bleeding, or use of any blood product transfusion.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 5.1 | 8.5
Statistical Analysis 1: Comparison: Bivalirudin vs Standard of Care: Heparins With Optional GPI; Test type: Superiority or Other; p = 0.0014, Chi-squared; Relative risk = 0.60, 95% CI 2-sided [0.43 to 0.82]

2. Secondary Outcome: The Composite Incidence of Death, Re-infarction (MI), or Non-CABG Major Bleeding
Description: A participant had a composite event if the participant experienced at least 1 of the 3 components (death, re-infarction [MI], or non-CABG major bleeding) of the composite. Incidence=the number of participants to experience the event/total number of at risk participants x 100. Death was defined as death from any cause at any time. Non-CABG major bleeding was defined as any one of the following: intracranial, retroperitoneal, intraocular, access site hemorrhage requiring radiological or surgical intervention, reduction in Hb concentration of >4 g/dL without an overt source of bleeding, reduction in hemoglobin concentration of >3 g/dL with an overt source of bleeding, re-intervention for bleeding, use of any blood product transfusion. MI was defined as a positive diagnosis of re-infarction (new event) not associated with index PCI.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 6.6 | 9.2

3. Secondary Outcome: The Incidence of Death, Re-infarction, Non-CABG-related Major Bleeding, or Ischemia-driven Revascularization (IDR)
Description: Incidence=number of participants to experience the event/total number of at risk participants x 100. Death from any cause at any time. Re-infarction was a positive diagnosis of re-infarction not associated with index PCI. Non-CABG major bleeding was any 1 of: intracranial, retroperitoneal, intraocular, access site hemorrhage requiring radiological or surgical intervention, reduction in Hb concentration of >4 g/dL without an overt source of bleeding, reduction in hemoglobin concentration of >3 g/dL with an overt source of bleeding, re-intervention for bleeding, use of any blood product transfusion. IDR was any refractory ischemia-driven repeat percutaneous intervention or bypass graft surgery involving any native coronary or pre-existing bypass graft vessel. In the absence of pain, new ST segment changes indicative of ischemia, acute pulmonary edema, ventricular arrhythmias, or hemodynamic instability presumed to be ischemic in origin, will constitute sufficient evidence of ischemia.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants
  Death | 2.9 | 3.1
  Re-infarction | 1.7 | 0.9
  Non-CABG-related major bleeding | 2.6 | 6.0
  IDR | 2.2 | 1.5

4. Secondary Outcome: The Incidence of Death at 1 Year
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Death was defined as death from any cause at any time.
Time Frame: Within 1 Year
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 5.4 | 5.3

5. Secondary Outcome: The Incidence of Major Bleeding: Thrombolysis in MI (TIMI) and Global Utilization of Streptokinase and tPA for Occluded Coronary Arteries (GUSTO)
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Major bleeding based on TIMI criteria was defined as any intra-cranial bleeding, or any bleeding associated with clinically overt signs associated with a drop in Hb of >5 g/dL (or, when Hb was not available, an absolute drop in hematocrit [Hct] >15%). Major bleeding based on GUSTO criteria was defined as severe/life-threatening: intra-cranial hemorrhage or resulting in substantial hemodynamic compromise requiring treatment.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants
  Major bleeding: TIMI | 1.3 | 2.1
  Major bleeding: GUSTO | 1.3 | 2.3

6. Secondary Outcome: The Incidence of Minor Bleeding: TIMI and GUSTO
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Minor bleeding based on TIMI criteria was defined as any clinically overt sign of bleeding (including observation by imaging techniques) that was associated with a fall in Hb of ≥3 g/dL and ≤5 g/dL (or, when Hb was not available, an absolute drop in Hct of ≥9% and ≤15%). Minor bleeding based on GUSTO criteria was defined as other bleed not requiring blood transfusion or causing hemodynamic compromise.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants
  Minor bleeding: TIMI | 6.5 | 11.2
  Minor bleeding: GUSTO | 6.5 | 11.0

7. Secondary Outcome: The Incidence of Stent Thrombosis (Academic Research Consortium [ARC Definition])
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Stent thrombosis, based on the ARC definition, was defined as angiographic confirmation of stent thrombosis, non-occlusive thrombus, occlusive thrombus, or pathological confirmation of stent thrombosis.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 1.6 | 0.5

8. Secondary Outcome: The Incidence of Thrombocytopenia
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Thrombocytopenia was defined as a post-procedural platelet count <100,000 cells/millimeter cubed (cells/mm^3) in a participant with a baseline or pre-procedural platelet count >100,000 cells/mm^3.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 0.7 | 1.4

9. Secondary Outcome: The Incidence of Stroke
Description: Incidence=the number of participants to experience the event/total number of at risk participants x 100. Stroke was defined as a sudden, focal neurological defect resulting from a cerebrovascular cause, resulting in death or lasting greater than 24 hours that was not due to a readily identifiable cause, such as a tumor, infection, or trauma.
Time Frame: Within 30 days
Population: Participants who were randomized and signed an ICF; ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Number analyzed (Participants) | 1089 | 1109
percentage of participants | 0.6 | 1.0

ADVERSE EVENTS:
Time Frame: From screening to Day 30
Arm/Group | Bivalirudin | Standard of Care: Heparins With Optional GPI
Serious Adverse Events (participants affected / at risk) | 145/1099 | 129/1094
Other Adverse Events (participants affected / at risk) | 134/1099 | 119/1094
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=1099) | Standard of Care: Heparins With Optional GPI (N=1094)
Ventricular fibrillation (Cardiac disorders) | 39 | 28
Cardiogenic shock (Cardiac disorders) | 21 | 17
Cardiac arrest (Cardiac disorders) | 7 | 17
Cardiac failure (Cardiac disorders) | 8 | 10
Coronary artery dissection (Cardiac disorders) | 7 | 2
Ventricular tachycardia (Cardiac disorders) | 3 | 4
Bradycardia (Cardiac disorders) | 2 | 3
Atrioventricular block complete (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 2 | 3
Intracardiac thrombus (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Coronary artery perforation (Cardiac disorders) | 2 | 1
Ventricular septal defect acquired (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Coronary no-reflow phenomenon (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricle rupture (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Papillary muscle rupture (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Interventricular septum rupture (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac asthma (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 5 | 3
Multi-organ failure (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 5
Septic shock (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriogram coronary (Investigations) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 4
Renal failure (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 2 | 0
Reperfusion injury (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=1099) | Standard of Care: Heparins With Optional GPI (N=1094)
Ventricular tachycardia (Cardiac disorders) | 57 | 39
Atrial fibrillation (Cardiac disorders) | 35 | 35
Bradycardia (Cardiac disorders) | 20 | 25
Hypotension (Vascular disorders) | 22 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days